CLINICAL TRIAL: NCT04197024
Title: Evaluation of the Impact of Immersive Virtual Reality During the Submaximal Cardiorespiratory Fitness
Brief Title: Assessment of Exercise Capacity in Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Opole University of Technology (Other)
Responsible Party: Principal Investigator, Sebastian Rutkowski, Principal Investigator, The Opole University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: OpoleUofTech1
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers
Keywords: virtual reality; COPD; exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Each individual will be evaluated by a traditional test and a virtual reality test.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional exercise capacity test (Experimental): Patients of the Ministry of the Interior and Administration hospital in Głuchołazy with a diagnosed disease unit of Chronic Obstructive Pulmonary Disease (COPD).
  Interventions: Device: Exercise capacity test; Device: Exercise capacity test in virtual reality
- Immersive virtual reality exercise capacity test (Experimental): Healthy volunteers, Students of Department of Physical Education and Physiotherapy, Opole University of Technology, Opole, Poland
  Interventions: Device: Exercise capacity test; Device: Exercise capacity test in virtual reality

INTERVENTIONS:
Device: Exercise capacity test — Patients will be assessed by symptom-limited maximal cardiopulmonary exercise testing (CPET) following a 25W, tree-minute stage, beginning at 25W (healthy volunteers will start the test with a load of 50W). For both sexes and arms, participants will be instructed during the test to remain at the frequency between 60 to 80 rotations per minute (rpm). Heart rate (HR) will be continuously recorded using a monitor Polar H10.
  Other Names: Cardiopulmonary Exercise Testing
Device: Exercise capacity test in virtual reality — Patients will be assessed by symptom-limited maximal cardiopulmonary exercise testing (CPET) following a 25W, tree-minute stage, beginning at 25W (healthy volunteers will start the test with a load of 50W). For both sexes and arms, participants will be instructed during the test to remain at the frequency between 60 to 80 rotations per minute (rpm).Heart rate (HR) will be continuously recorded using a monitor Polar H10. VR HTC Vive Pro goggles along with VR health care (aerobic exercise) VR Cycling software will be used for stimulation throughout the duration of the test. The HTC Vive Tracker device will be also use to link images in virtual reality with the pedal speed.
  Other Names: Cardiopulmonary Exercise Testing in virtual reality

SUMMARY:
The 20th century brought a dynamic development of new technologies, including virtual reality (VR). VR is an artificial image generated by IT technologies. It is most often associated with entertainment, but has a much wider application in other fields. The aim of the study is to assess the influence of the application of immersive virtual reality during an exercise capacity test on a bicycle ergometer.

DETAILED DESCRIPTION:
Scientists suggests that there are four types of virtual reality: immersive virtual reality, desktop virtual reality (i.e., low-cost homebrew virtual reality), projection virtual reality, and simulation virtual reality. The sense of presence or immersion is a critical feature distinguishing virtual reality from other types of computer applications. It seems interesting whether immersion in virtual reality can influence the assessment of exercise capacity. The aim of the study is to assess the influence of the application of immersive virtual reality during an exercise capacity test on a bicycle ergometer. It is assumed that an exercise capacity test on a cycloergometer will be performed in a traditional form and in a virtual reality.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male, age: 20-25 years

Exclusion Criteria:

1. diagnosed internal diseases
2. diseases and injuries of the locomotors system impairing the function of transport 3 Cognitive disorders preventing contact with the patient, Mini-Mental State Examination < 24 points.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Exercise Testing- cycle ergometer | First or second day of the assessment - the traditional exercise test
  The exercise test on an electronically-braked cycle ergometer (Lode Excalibur Sport PFM) was used for evaluation. Test began with a unloaded cycling for 3 minutes, then 50W for 3 minutes followed by an incremental phase in which work rate increased by 25 watts every 3 minutes. Heart rate (HR) was continuously recorded. These submaximal tests were terminated when the subjects reached 85% of the age-predicted maximal HR (calculated as 220 - age)
HRV | First or second day of the assessment - the exercise test in VR
  The Polar H10 monitor (Polar Electro Oy Inc., Kempele, Finland) was employed to record heart rate series at a sampling frequency of 1000 Hz. All HRV analyses were carried out with the Kubios HRV Premium version 3.3.1 (HRV analysis, University of Eastern Finland). The R-R interval series were filtered with the artifact correction algorithm which was set at the automatic mode. Time- and frequency-domain HRV parameters were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Rutkowski, PhD, Principal Investigator — The Opole University of Technology
Locations (1):
- Institute of Physiotherapy, Department of Physical Education and Physiotherapy, Opole University of Technology, Opole, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutkowski S, Szary P, Sacha J, Casaburi R. Immersive Virtual Reality Influences Physiologic Responses to Submaximal Exercise: A Randomized, Crossover Trial. Front Physiol. 2021 Sep 30;12:702266. doi: 10.3389/fphys.2021.702266. eCollection 2021. PMID 34658904